CLINICAL TRIAL: NCT07405047
Title: Fractionated Stereotactic Radiotherapy for Limited Small Brain metastases--a Phase II Trial
Brief Title: Fractionated Stereotactic Radiotherapy for Limited Small Volume Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, YE ZHANG, Dr., Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-012829
Record Dates: First submitted 2024-05-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Brain Metastases, Adult
Keywords: limited brain metastases; small brain metastases; fractionated stereotactic radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fractionated stereotactic radiotherapy group (Experimental): fractionated stereotactic radiotherapy is given to all the patients. The presciption is 30 Gy in 5 fractions.
  Interventions: Radiation: fractionated stereotactic radiotherapy

INTERVENTIONS:
Radiation: fractionated stereotactic radiotherapy — The prescription is 30 Gy in 5 fractions.

SUMMARY:
This is a single-center, open lable, single-arm phase II clinical study to evaluate the efficacy and safety of fractionated stereotactic radiotherapy (FSRT) in patients with 1-4 brain metastases with ≤2cm in diameter.

DETAILED DESCRIPTION:
This study plans to enroll 48 patients with 1-4 brain metastases with ≤2cm in diameter. All of the patients will receive FSRT with the dose of 30 Gy in 5 fractions. The primary endpoint is local control rate of asymptomatic brain necrosis at 1 year. The secondary endpoints include disease control rate at 2 months, local control rate at 1 year, intra-cranial distant failure at 1 year, overall survival rate at 1 year, toxicities, radiation necrosis rate, etc.

ELIGIBILITY:
Inclusion Criteria:

1. The primary tumor is proved malignant by pathology;
2. Brain metastases are confirmed by enhanced MRI, and the number of lesions is 1-4;
3. The maximum diameter of each lesion is ≤ 2cm;
4. Age ≥ 18 years old;
5. KPS≥ 70;
6. Brain metastases haven't been previously treated locally and patients haven't received prior whole brain radiotherapy (WBRT);
7. expected survival of more than 6 months;
8. The functions of vital organs meet the requirements;
9. The patients voluntarily join the clinical study and sign the informed consent.

Exclusion Criteria:

1. Surgical intervention is considered for MDT consultation;
2. Meningeal metastasis;
3. The primary tumor is small cell lung cancer;
4. Follow-up data can't be obtained regularly;
5. patients are combined with other serious diseases, such as serious cardiovascular diseases: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including QTc interval ≥ 450 ms in men and ≥ 470 ms in women); Patients with grade Ⅲ to Ⅳ cardiac insufficiency or left ventricular ejection fraction (LVEF) < 50% indicated by color doppler examination;
6. neurological lesions such as cerebral hemorrhage and cerebral infarction occurred within 6 months;
7. Other circumstances that, in the investigator's judgment, would render the subject unfit for study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
local control without symptomatic radiation necrosis rate | 1 year after fractionated stereotactic radiotherapy (FSRT)
  radiation necrosis (RN) is defined as: enhanced MRI after radiotherapy shows lace or irregular enhancement around the lesion, less enhancement in the center of T1-WI, high signal around the lesion of T2-WI, and no nodules of equal intensity or low intensity, and no obvious diffusion restriction in DWI sequences. RN can be diagnosed if the above brain MRI findings still exist after 3 months of re-xamination.

SECONDARY OUTCOMES:
disease control rate | 2 months after fractionated stereotactic radiotherapy (FSRT)
  Complete release (CR) + partial release (PR) + stable disease (SD) rate, assessed by RECIST 1.1 criteria
local control rate | 1 year after fractionated stereotactic radiotherapy (FSRT)
  local control rate of the lesions which received FSRT
intra-cranial distant failure rate | 1 year after fractionated stereotactic radiotherapy (FSRT)
  new brain metastases in the brain
intra-cranial progression free survival rate | 1 year after fractionated stereotactic radiotherapy (FSRT)
  local control without intra-cranial distant failure
adverse events | From date of fractionated stereotactic radiotherapy (FSRT) until the date of first documented progression, assessed up to 36 months.
  neurological toxicity was determined according to RTOG acute toxicity classification criteria, and the rest was determined according to NCI-CTCAE V5.0 criteria
radiation necrosis rate | From date of fractionated stereotactic radiotherapy (FSRT) until the date of first documented progression, assessed up to 36 months.
  radiation necrosis (RN) is defined as: enhanced MRI after radiotherapy shows lace or irregular enhancement around the lesion, less enhancement in the center of T1-WI, high signal around the lesion of T2-WI, and no nodules of equal intensity or low intensity, and no obvious diffusion restriction in DWI sequences. RN can be diagnosed if the above brain MRI findings still exist after 3 months of re-xamination.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Zhang, MD., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Ye Zhang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD is protected by our institution and are not allowed to share to others.